CLINICAL TRIAL: NCT06467565
Title: A Phase II Study of Liposomal Irinotecan (Nal-IRI) With 5 Fluorouracil, Leucovorin, and Oxaliplatin (NALIRIFOX) in Patients With Locally Advanced Pancreatic Cancer
Brief Title: NALIRIFOX as Induction Therapy in LAPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Kuirong Jiang, Pro, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-254
Record Dates: First submitted 2024-06-15; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NALIRIFOX (Experimental): NALIRIFOX（Oxaliplatin 60 mg/m2 IV over 2 hours ; Liposomal Irinotecan 50 mg/m2 IV over 90 minutes ; Leucovorin(l-LV) 400 mg/m2 IV over 2 hours 5-fluorouracil 2.4 g/m2 for 46 hours continuous infusion） on days 1 of a 14-day cycle.
  Interventions: Drug: Liposomal irinotecan

INTERVENTIONS:
Drug: Liposomal irinotecan — NALIRIFOX（Oxaliplatin 60 mg/m2 IV over 2 hours ; Liposomal Irinotecan 50 mg/m2 IV over 90 minutes ; Leucovorin(l-LV) 400 mg/m2 IV over 2 hours 5-fluorouracil 2.4 g/m2 for 46 hours continuous infusion） on days 1 of a 14-day cycle.

SUMMARY:
This is a prospective, single arm, single center, phase II study of NALIRIFOX as conversion therapy in patients with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
Subjects will be treated with the NALIRIFOX regimen every 2 weeks in 4-weeks cycles Imaging of tumor lesions will be performed after the subject has completed the first 2 cycles of treatment, and if the subject has not progressed, the subject will continue treatment until surgical resection, disease progression (RECIST 1.1) or intolerable toxicity, start of new anticancer drug therapy, withdrawal from the study, death, or loss to follow-up. All treated subjects will be evaluated for response while on this treatment every 8 weeks (±7) days after until surgical resection, disease progression (RECIST 1.1), intolerable toxicity, start of new anticancer drug therapy, withdrawal from the study, death, or loss to follow-up.. After 24 weeks of treatment, capecitabine or S-1 is the maintenance regimen. Radiographic response will be evaluated every 12 weeks (± 7 days) during the maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, ≤ 70 years old, male or female;
2. Understand the objectives and benefits and risks of the clinical trial, voluntarily participate in and sign the informed consent form;
3. ECOG score 0-1;
4. The subject had histopathologically or cytologically confirmed type of pancreatic ductal adenocarcinoma
5. Local progression according to the 2022 CSCO guidelines;
6. Initial subjects with locally advanced pancreatic cancer who have not undergone resection of pancreatic tumor (except open exploration or internal drainage surgery), chemotherapy, targeted, or immunotherapy.
7. At least one measurable pancreatic lesion per RECIST 1.1 criteria;
8. Expected survival time ≥ 3 months.
9. Heart, lung, liver, kidney and other major organ functions are basically normal.
10. Hematology tests should meet the following criteria (no blood transfusion, no use of blood products, granulocyte colony-stimulating factor, or other hematopoietic growth factors within 7 days prior to hematology):

    1. White blood cell count ≥ 3.0 × 109/L and neutrophil count ≥ 1.5 × 109/L.
    2. Platelet count ≥ 100 × 109/L.
    3. Hemoglobin ≥ 90 g/L.
    4. If component blood transfusions (red blood cells, platelets, etc.) are received at screening, reexamination of hematology must be performed at 1-week intervals before further screening can be considered.
11. Blood chemistry tests should meet the following criteria:

    1. Plasma total bilirubin ≤ 1.5 × upper limit of normal.
    2. ALT, AST, or ALP ≤ 2.5 × upper limit of normal;
    3. Creatinine clearance ≥30 mL/min calculated by the Cockcroft-Gault formula (Cockcroft-Gault formula: male Ccr = [(140-age) × body weight (kg)]/[0.818 × Scr (μmol/L)] or Ccr = (140-age) × body weight (kg)/72 × Scr (mg/dl), and female Ccr calculated as male × 0.85);
12. The subject had no symptoms of cardiac insufficiency (NYHA functional class ≤ II) at baseline and had no obvious abnormalities or abnormalities in electrocardiograms that were not clinically significant.
13. Good compliance, voluntary compliance with this clinical trial protocol and follow-up by the investigator during the study.
14. Subjects of childbearing potential voluntarily take highly effective contraceptive measures in the trial.
15. Females must be non-lactating.

Exclusion Criteria:

1. Known allergy or intolerance to the ingredients or excipients of this investigational product.
2. Any metastatic lesions.
3. Patients with unresolved acute or chronic infection
4. Other malignancies within 5 years (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
5. Active hepatitis.
6. Patients with portal hypertension or cavernous transformation of the portal vein; patients with gastrointestinal bleeding caused by tumor involving the digestive tract; patients with intra-abdominal fistula or abscess due to tumor involvement of digestive tract; the tumor encircles the celiac trunk or SMA and causes significant vascular wall involvement (worm-like changes);
7. Presence of third space effusion that cannot be controlled by drainage or other means (e.g., moderate-large pleural effusion, moderate-large pericardial effusion, ascites); a small amount of pleural effusion or ascites that is not clinically symptomatic and does not require clinical intervention should be strictly controlled before enrollment.
8. Mental illness or mental disorder, poor compliance, unable to cooperate with treatment
9. Patients with severe organic diseases or major organ failure, such as decompensated heart and lung failure, which lead to intolerance to chemotherapy.
10. Abnormal coagulation (INR > 1.5, APTT > 1.5 ULN), bleeding tendency (e.g., active ulcer lesions in the stomach, occult blood in stool (+ +), melena and/or hematemesis within 3 months, hemoptysis) or near the location of the lesion to major vessels.
11. Patients with Grade I or higher coronary heart disease, arrhythmia (including QTc prolongation > 450 ms in males and > 470 ms in females), taking arrhythmic drugs, or associated underlying heart disease and cardiac insufficiency.
12. Patients with renal insufficiency, previous renal disease, and positive urine protein (urine protein test 2 + or more, or 24-hour urineprotein quantitation > 1.0 g).
13. Organ transplant recipients.
14. There are drug addicts and other adverse drug addicts, long-term alcoholics and AIDS and other infectious diseases.
15. Long-term use of corticosteroids or immunosuppressants.
16. Those who have received vaccines (including live and live attenuated vaccines) within 4 weeks prior to enrollment, such as measles, mumps, rubella, varicella, yellow fever, rabies, BCG, and typhoid (oral) vaccines, etc., or who plan to be vaccinated during study dosing; Allowing all types of COVID-19 vaccines.
17. Subjects with active hepatitis B or hepatitis C (HBV DNA ≥ 1 × 104 copies or ≥ 2000 IU/mL regardless of drug control; hepatitis C infection, HCV RNA ≥ 15 IU/mL); or HIV antibody positive (testing is not required if there is no clinical evidence of possible HIV infection); or syphilis antibody (TPPA) positive.
18. Breast feeding, known pregnancy, positive serum pregnancy test or unwillingness to use a reliable method of birth control, during therapy and for 6 months following the last dose of nal-IRI. Females of Childbearing Potential must either agree to use and be able to take effective contraceptive birth control measures (Pearl Index < 1) or agree to use effective contraception during treatment and for at least 7 months after last application of program treatment. Males with female partners of reproductive potential should use condoms during treatment and for 4 months after the last dose. A female subject is considered to be of childbearing potential unless she is age ≥ 50 years and naturally amenorrhoeic for ≥ 2 years, or unless she is surgically sterile. Males must agree not to father a child (including not donating sperm) during the course of the trial and for at least 6 months after last administration of study drugs.
19. In the opinion of the investigator, the subject is unable to complete the entire trial process or other circumstances that are not suitable for participation in this trial.
20. Use of strong inhibitors or inducers of CYP3A, CYP2C8 and UGT1A1. Subjects are ineligible if:

    * they are unable to discontinue the use of strong inhibitors of CYP3A, CYP2C8 and UGT1A1 at least 1 week prior to first dosing
    * they are unable to discontinue the use of strong CYP3A and CYP2C8 inducers at least 2 weeks prior to first dosing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 1 year
  ORR is defined as the percentage of participants who have a confirmed complete response or partial response according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to two years
  PFS is defined as the time from enrollment of the trial to the first documented disease progression or death due to any cause.
Overall survival (OS) | Up to two years
  The duration from the date of recruitment to the date of death from any cause.
Adverse events (safety) | Up to two years
  Adverse events (safety ) will be evaluated according to the NCI CTCAE Version 5.0.The number and severity of treatment-related side effects, including AE and SAE, will be recorded during treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided